CLINICAL TRIAL: NCT02700971
Title: Rational Approach To Immuno-Oncology Microarray Prediction of Response to Nivolumab, Ipilimumab, or Combined Therapy in Subjects With Previously Untreated, Locally Advanced or Metastatic Melanoma
Brief Title: RATIO: Rational Approach To Immuno-Oncology
Acronym: RATIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Transplant Genomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IIT-RATIO-CCI-01
Record Dates: First submitted 2016-02-29; First posted 2016-03-07 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cutaneous Biopsy for microarray analysis (Experimental): To determine whether outcomes improve as a function of anti-tumor immunity which may enable the use of this technique as a predictive biomarker of treatment response.
  Interventions: Procedure: Molecular Microscope Diagnostic system

INTERVENTIONS:
Procedure: Molecular Microscope Diagnostic system — Consented patients with locally advanced or metastatic melanoma with This trial will utilize a Molecular MicroscopeTM diagnostic system (MMDxTM) that combines the molecular and histopathological features of biopsies, plus clinical and laboratory parameters, to create the first Integrated Diagnostic System. This MMDxTM will be utilized to phenotype cutaneous melanoma biopsy samples to detect an immune responsive mRNA signature.

SUMMARY:
This trial will utilize a Molecular MicroscopeTM diagnostic system (MMDxTM) that combines the molecular and histopathological features of biopsies, plus clinical and laboratory parameters, to create the first Integrated Diagnostic System. This MMDxTM will be utilized to phenotype cutaneous melanoma biopsy samples to detect an immune responsive mRNA signature.

DETAILED DESCRIPTION:
The trial treatment will consist of a pretreatment 18 gauge core biopsy of locally advanced or metastatic cutaneous or subcutaneous lesions. The biopsies will be stabilized on site in RNAlater and shipped to ATAGC by courier at ambient temperature. RNA will be extracted using Trizol-chloroform method and purified using RNAEasy micro kit (Qiagen). RNA samples passing the quality control test (Agilent Bioanalyzer) will be labeled, hybridized to PrimeView Affymetrix microarrays and scanned according to the manufacturer's protocol. Resulting ".CEL" files will be used for the analysis of the global gene expression.

Pathogenesis Based Transcript (PBT) sets that represent molecular signatures of inflammation will be assessed in core biopsies from melanoma patients. Each PBT set gets a "score" - a summarized expression of all members of a set. PBT scores allow an estimate of pre and post-treatment immunological activity in each tumor e.g. TCMR activity or macrophage burden. PBT scores will be correlated with clinical outcome to determine the utility of this technology as a prognostic and predictive biomarker. Finally a molecular classifier predicting the response to therapy will be built.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, > 18 years of age
* Histologically confirmed locally advanced or metastatic melanoma with cutaneous or subcutaneous lesions
* Immunotherapy treatment naïve subjects (ie, no prior systemic anticancer therapy for unresectable or metastatic melanoma)
* Scheduled to receive ipilimumab, nivolumab, or combination treatment
* Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2
* Not pregnant or lactating. Women who are of child-bearing potential must agree to use an effective means of birth control (i.e., latex condom, diaphragm, cervical cap, etc) to avoid pregnancy.
* Informed consent for microarray analysis of locally advanced lesion or skin metastasis retrieved by standard of care biopsy

Exclusion Criteria:

* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co- stimulation or immune checkpoint pathways
* Subjects with active, known, or suspected autoimmune disease
* If considered high-risk and tested for hepatitis: Any positive test result for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Any significant medical condition, laboratory abnormality, or psychiatric illness, that would prevent the subject from participating in the study, places the subject at unacceptable risk if he/she were to participate in the study, or any condition that confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Correlation of the MMDx from pretreatment biopsy with overall response rate (ORR). | 24 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
Overall Survival (OS) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Smylie, MB, FRCPC, Principal Investigator — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No